CLINICAL TRIAL: NCT00516607
Title: Phase I Study of Enzastaurin and Temozolomide in Patients With Gliomas
Brief Title: Enzastaurin and Temozolomide in Treating Patients With Primary Gliomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26054; EORTC-26054
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult mixed glioma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult anaplastic ependymoma; adult giant cell glioblastoma; adult gliosarcoma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma; Ependymoma; Gliosarcoma | interventions — Temozolomide

INTERVENTIONS:
Drug: enzastaurin hydrochloride
Drug: temozolomide
Other: pharmacological study

SUMMARY:
RATIONALE: Enzastaurin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving enzastaurin together with temozolomide may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of enzastaurin when given together with temozolomide in treating patients with primary gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess if full doses of enzastaurin hydrochloride and temozolomide can be used in combination for the treatment of patients with primary gliomas.
* To determine the recommended phase II dose.

OUTLINE: This is a multicenter study.

Patients receive oral enzastaurin hydrochloride once or twice daily on days 1-28* and oral temozolomide once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *During the first course only, patients also receive enzastaurin hydrochloride on day -1.

Patients undergo blood sample collection on day 22 of course 1 and on day 5 of course 2 for pharmacokinetic studies of enzastaurin hydrochloride.

After completion of study treatment, patients are followed within 30 days and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary supratentorial glioma

  * WHO histologic grade 3 or 4

    * Patients who have undergone prior treatment for low-grade glioma that has transformed to glioblastoma (biopsy proven) allowed
* Amenable to standard temozolomide treatment
* First or second recurrent disease after prior surgery and/or radiotherapy OR newly diagnosed disease that is not amenable to radiotherapy (e.g., multifocal disease)

PATIENT CHARACTERISTICS:

* ECOG or WHO performance status 0-2
* Hemoglobin ≥ 10.0 g/dL
* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase and transaminases ≤ 2.5 x ULN
* Serum creatinine < 1.7 mg/dL
* Not pregnant or lactating
* Negative pregnancy test
* Fertile patients must use effective contraception
* Clinically normal cardiac function
* No ischemic heart disease within the past 6 months
* No clinically significant abnormalities or uncontrolled cardiac arrhythmia by ECG
* QTc interval ≤ 450 msec (males) or ≤ 470 msec (females) by baseline 12-lead ECG
* No history of congenital long QTc syndrome
* No history of stroke
* No other prior or concurrent malignancy within the past 5 years except cone biopsied carcinoma of the cervix or adequately treated basal or squamous cell skin carcinoma
* No unstable systemic diseases
* No active uncontrolled infections
* No uncontrolled hypertension
* No psychological, familial, sociological, or geographical condition that would preclude study participation
* Must be able to swallow tablets

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 1 prior chemotherapy regimen in the adjuvant setting or for first recurrence
* Prior temozolomide allowed provided there was no disease progression during temozolomide treatment or within 6 weeks of completing temozolomide treatment
* Prior surgery for primary brain tumor within the past 3 months allowed
* Patients who are receiving corticosteroid treatment must be on a stable or decreasing dose for at least 1 week before study entry
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 14 days since prior and no concurrent enzyme-inducing antiepileptic drugs including, but not limited to, any of the following:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
* More than 30 days since prior and no other concurrent investigational treatments
* No concurrent anticoagulant treatment (e.g., warfarin)

  * Low molecular weight heparin for patients who require anticoagulant therapy after starting study treatment may be allowed
* No concurrent routine use of colony-stimulating factors
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose
Dose-limiting toxicity

SECONDARY OUTCOMES:
Response rate
Progression-free survival
Overall survival
Pharmacokinetics of enzastaurin hydrochloride alone and in combination with temozolomide

CONTACTS AND LOCATIONS:
Overall Officials: Roy Rampling, MD, PhD, Study Chair — University of Glasgow
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Rampling R, Sanson M, Gorlia T, Lacombe D, Lai C, Gharib M, Taal W, Stoffregen C, Decker R, van den Bent MJ. A phase I study of LY317615 (enzastaurin) and temozolomide in patients with gliomas (EORTC trial 26054). Neuro Oncol. 2012 Mar;14(3):344-50. doi: 10.1093/neuonc/nor221. Epub 2012 Jan 29. PMID 22291006